CLINICAL TRIAL: NCT02200848
Title: A Phase I Study of Lenalidomide in Combination With Rituximab and Ibrutinib in Relapsed and Refractory CLL and SLL
Brief Title: Phase I Study of Lenalidomide, Rituximab and Ibrutinib in Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recruitment difficulties and toxicity
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI#9540
Record Dates: First submitted 2014-07-22; First posted 2014-07-25 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2017-05

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Lenalidomide; Ibrutinib; Rituximab; CLL; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; ibrutinib; Rituximab; glutarimide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide, Ibrutinib, Rituximab (Experimental): Rituximab on day 1, lenalidomide days 1-21 and ibrutinib continuously for 6 cycles or until disease progression or intolerance to the combination. Single agent ibrutinib will then be continued until disease progression or intolerance.
  Interventions: Drug: Lenalidomide, Ibrutinib, Rituximab

INTERVENTIONS:
Drug: Lenalidomide, Ibrutinib, Rituximab — Dose level -2 Ibrutinib 280 mg; Lenalidomide 2.5 mg; Rituximab 375 mg/m2 Level -1 Ibrutinib 420 mg; Lenalidomide 2.5 mg; Rituximab 375 mg/m2 Level 1 Ibrutinib 420 mg; Lenalidomide 5 mg; Rituximab 375 mg/m2 Level 2 Ibrutinib 420 mg; Lenalidomide 10 mg; Rituximab 375 mg/m2 Level 3 Ibrutinib 420 mg; Lenalidomide 15 mg; Rituximab 375 mg/m2
  Other Names: Ibrutinib; PCI-32765; NSC# 748645; Imbruvica; Lenalidomide; alpha-[3-aminophthalimido] glutarimide; Revlimid; CC-5013; NSC#703813; Rituximab; IDEC-C2B8; Rituxan

SUMMARY:
This study is for subjects diagnosed with recurrent or relapsed CLL/SLL. The purpose of this study is to test the safety of the combination of the drugs lenalidomide and ibrutinib at different dose levels, in combination with the drug rituximab. We want to find out what effects, good and/or bad, they have on patients with CLL/SLL.

The hypothesis of the study is that it will be safe to give the three drugs in combination and the information learned from this trial will be used to study the 3 drug combination is a larger future trial.

DETAILED DESCRIPTION:
Treatment consists of dose escalations of lenalidomide and ibrutinib and fixed doses of rituximab. A small expansion cohort to include 10 patients will follow once the recommended phase II dose is found.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated chronic lymphocytic leukemia or small lymphocytic lymphoma that requires treatment
* No prior systemic treatment within 4 weeks of enrollment
* No corticosteroids within 2 weeks prior to study entry
* Measurable disease must be present
* No concomitant anti-cancer therapies
* ECOG status </= 2
* Patients with HIV infection are eligible
* Patients with treated CLL or SLL in CNS are eligible
* Non-pregnant and non-nursing
* Life expectancy greater than 60 days
* Adequate bone marrow, kidney and liver function
* No major surgery within 28 days or minor surgery within 5 days of starting treatment

Exclusion Criteria:

* History od Richter's transformation
* History of prior allogeneic transplant
* Radioimmunotherapy within 1 year of enrollment
* Prior Bruton's tyrosine kinase inhibitor or lenalidomide
* History of allergic reactions to compounds similar to ibrutinib, lenalidomide or rituximab or hypersensitivity
* active or uncontrolled autoimmune hemolytic anemia or ITP
* Transfusion-dependent thrombocytopenia or bleeding disorders
* Active hepatitis B or C infections
* History of known Human Anti-Chimeric Antibody positivity
* History of erythema multiforme, toxic epidermal necrolysis, or Stevens-Johnson syndrome
* History of uncontrolled seizures
* Autoimmune disorder that requires active immunosuppression
* Stroke or intracranial hemorrhage within last 6 months
* History of congestive heart failure, myocardial infarction, unstable angina, uncontrolled arrhythmia or any Class 3 or 4 heart disease in the last 6 months
* No prior malignancy except if treated with curative intent with no active disease for more than 3 years; adequately treated non-melanoma skin cancer or cervical cancer in situ
* using warfarin or similar Vitamin K antagonists Unable to swallow capsules or disease significantly affecting gastrointestinal function or inhibiting small intestine absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-04; Primary Completion 2017-03-27 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Recommended Phase II dose | 1year
  The dose at which less than 2 of 6 patients experience a dose limiting toxicity

SECONDARY OUTCOMES:
Safety | 2 years
  adverse events, serious adverse events, adverse events leading to discontinuation, deaths
Antitumor efficacy | 2 years
  Proportion of patients who achieve stable disease, partial or complete response; progression-free survival defined as duration of time from start of treatment to time of progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Chaitra Ujjani, MD, Principal Investigator — Georgetown Lombardi Comprehsnive Cancer Center
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Ujjani C, Wang H, Skarbnik A, Trivedi N, Ramzi P, Khan N, Cheson BD. A phase 1 study of lenalidomide and ibrutinib in combination with rituximab in relapsed and refractory CLL. Blood Adv. 2018 Apr 10;2(7):762-768. doi: 10.1182/bloodadvances.2017015263. PMID 29610115